CLINICAL TRIAL: NCT05158036
Title: Comparison of the Effects of Different Massage Techniques in Women With Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, associate professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/12/01
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classic massage group (Active Comparator): Classical massage will be applied to the lumbal and abdominal region 5 days a week, from the estimated date of ovulation until the next menstrual bleeding begins. The application will take approximately 15 minutes. During the massage, the physiotherapist will apply stroking and kneading movements by using baby oil. During the treatment of the lumbal region, the patient will be in the prone position; during the treatment of the abdominal region, the patient will be in the supine position.
  Interventions: Other: Classic massage group
- Connective tissue massage group (Active Comparator): Connective tissue massage will be applied to the lumbosacral, lower thoracic, abdominal and anterior pelvic regions 5 days a week, from the estimated date of ovulation until the onset of the next menstrual bleeding. The application will take approximately 15 minutes. During the massage, the physiotherapist will bring the tip of the middle finger of the hand into contact with the patient's skin and apply traction to the skin. During the treatment of the lumbar region, the patient will be in the sitting position, during the treatment of the abdominal and anterior pelvic region, the patient will be in the supine position.
  Interventions: Other: Connective tissue masage

INTERVENTIONS:
Other: Classic massage group — Classic massage application will be given to the Classic massage group
  Arms: Classic massage group
Other: Connective tissue masage — Connective tissue masage application will be given to the Connective tissue masage group
  Arms: Connective tissue massage group

SUMMARY:
The aim of this study was to compare the effects of different massage techniques on pain, primary dysmenorrhea (PD)-related symptoms and functional and emotional influence in women with PD.

DETAILED DESCRIPTION:
Primary dysmenorrhea is defined as painful menstrual cramps without an underlying pelvic pathology or organic problem. Massage, which is one of the physiotherapy methods that reduces pain by acting on the autonomic nervous system and circulation, has an important place in the management of PD among non-pharmacological treatment approaches. In the literature, there are studies on the use of classical massage and connective tissue massage in women with PD for reducing menstrual pain and PD-related symptoms. However, to the best of our knowledge, no study has been found comparing classical massage and connective tissue massage in PD management.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Women with a complaint of primary dysmenorrhea,
* Volunteer women who have a regular menstrual cycle (28 ± 7 days)
* Women who have menstrual pain intensity greater than 40 mm according to the Visual Analogue Scale considering the last 6 months

Exclusion Criteria:

* Having gastrointestinal, urogynecological, autoimmune, psychiatric diseases and/or other chronic pain syndromes,
* Those who have given birth,
* Those who have a pregnancy status,
* Those who use intrauterine devices,
* Those who have had pelvic surgery,
* Those who use chronic medications, including oral contraceptives or antidepressants, for at least 6 months before the study,
* Those with a pathological history and radiological findings showing secondary dysmenorrhea

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | change from baseline at an average of 2 weeks
  Menstrual pain intensity will be evaluated with Visual Analogue Scale.

SECONDARY OUTCOMES:
Pressure pain threshold | change from baseline at an average of 2 weeks
  Pressure pain threshold will be evaluated with algometer
Primary dysmenorrhea (PD)-related symptoms | change from baseline at an average of 2 weeks
  Severity of PD-related symptoms will be evaluated Visual Analogue Scale.
Functional and emotional effects | change from baseline at an average of 2 weeks
  Functional and emotional effects will be evaluated with Functional and Emotional Dysmenorrhea Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University